CLINICAL TRIAL: NCT05167110
Title: Nutritional Intervention in Children With ASD and/or ADHD: Randomized Controlled Trial With Probiotics.
Brief Title: Nutritional Intervention for Children With ASD and/or ADHD
Acronym: PRONED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Josefa Canals Sans, Professor, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UniversitatRoviraVirgili
Record Dates: First submitted 2021-12-20; First posted 2021-12-22 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: ADHD; ASD; Probiotics; Microbiota
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: ABBiotics has been the producer of probiotics and who knows the masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Children assigned to the groups (ASD/ADHD) will be randomly prescribed supplementation with two GABA- and dopamine-producing strains at a total of 1 x 10 (9) CFU/capsule for 12 weeks (probiotic subgroup).
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Children assigned to the groups (ASD/ADHD) will be randomly prescribed placebo supplementation for 12 weeks (placebo subgroup).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Children assigned to the groups (ASD/ADHD) will be randomly prescribed placebo supplementation for 12 weeks (placebo subgroup).
  Arms: Placebo group
Dietary Supplement: Probiotic — Children assigned to the groups (ASD/ADHD) will be randomly prescribed supplementation with two GABA- and dopamine-producing strains at a total of 1 x 10 (9) CFU/capsule for 12 weeks (probiotic subgroup).
  Arms: Treatment group

SUMMARY:
Based on alterations in the intestinal microbiota in children with ASD and the high comorbidity between ASD and ADHD, the aim of this project was to assess whether the administration of probiotics with strains related to the production of the neurotransmitters dopamine and GABA had a positive effect on social behavior, attention, and behavior.

DETAILED DESCRIPTION:
We hypothesized to find differences in the composition and / or function of the microbiota of the gastrointestinal tract of children with ASD and / or ADHD. We consider that the intervention with probiotics (and specifically with GABA and dopamine producing strains), can modify the composition and / or function of the GIT microbiota and change the child's behavior, partially reducing the symptoms of attention deficit, anxiety, irritability, impulsivity and restlessness associated with diagnoses and consequently, we believe that it could improve the quality of life for children and their families. Apart from the clinical evaluation of the disorder and associated psychopathological symptoms and neuropsychological deficit, the diet, lifestyle and anthropometric characteristics of the child will be evaluated, which can influence the composition and / or function of gut the microbiota.

The sample that will be part of the study will be 80 children, 40 with a diagnosis of ASD and 40 with a diagnosis of ADHD. These children will randomly receive placebo or probiotic intervention for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Parental informed consent,
* ASD and ADHD will meet the DSM diagnoses (edition IV-TR or 5) criteria
* Ages between 5 and 16 years
* To complete period (12weeks) of taking the probiotic

Exclusion Criteria:

* Having suffered adverse effects in the previous administration of probiotics
* Being on probiotics 3 months before the start of the intervention
* To suffer any medical illness incompatible with the administration of probiotics
* Having intolerances or allergies to the excipient of the treatment (probiotic or placebo)
* Taking antibiotics in the start of the intervention.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Continuous Performance Test (CPT 3 or CPT-K 2) | 12 weeks
  Measures attention and inhibitory control
Social Responsiveness Scale™, Second Edition | 12 weeks
  Assess severity of the ASD manifestations answered by parents
Conners scale | 12 weeks
  Assess severity ADHD symptoms answered by parents
Behavior Rating Inventory of Executive Function (BRIEF-2) | 12 weeks
  Assess severity ADHD symptoms answered by parents

SECONDARY OUTCOMES:
Physical Activity (PAQ-C) | 12 weeks
Gastrointestinal symptoms | 12 weeks
  Discomfort/abdominal lower pain
Child Behavior Checklist (CBCL) | 12 weeks
  emotional and behavioral symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Josefa Canals-Sans, MD, Principal Investigator — University Rovira i Virgili
Locations (1):
- University Rovira i Virgili, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Results

REFERENCES:
- [Derived] Rojo-Marticella M, Arija V, Canals-Sans J. Effect of Probiotics on the Symptomatology of Autism Spectrum Disorder and/or Attention Deficit/Hyperactivity Disorder in Children and Adolescents: Pilot Study. Res Child Adolesc Psychopathol. 2025 Feb;53(2):163-178. doi: 10.1007/s10802-024-01278-7. Epub 2025 Jan 11. PMID 39798036